CLINICAL TRIAL: NCT06240247
Title: Associations Between Birth Order, Sibship Size, Childhood Socioeconomic Factors, Perinatal Characteristics and Oral Health Related Quality of Life and Periodontal Disease
Brief Title: Associations Between Birth Order, Sibship Size and Periodontal Disease
Status: Completed | Type: Observational
Sponsor: Zeynep Tastan Eroglu (Other)
Responsible Party: Sponsor-Investigator, Zeynep Tastan Eroglu, Assistant professor, Necmettin Erbakan University
Organization: Necmettin Erbakan University (Other)
Other Study IDs: BirthOrder
Record Dates: First submitted 2024-01-22; First posted 2024-02-05 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gingival healthy: People who do not have clinical attachment loss in their gums, pocket or bone loss, and whose bleeding percentage in their gums is 10% or less
- Gingivitis: People who do not have clinical attachment loss in their gums, pocket or bone loss, and whose bleeding percentage in their gums is 10% or more

SUMMARY:
The goal of this observational study is to learn about the relationship between sibship size, birth order, gingival health, and oral health habits in systematical healthy participants. The main questions it aims to answer are:

question 1: Is there any association between birth order and gingival health? question 2: Is there any association between birth order and oral health habits? question 3: Is there any association between birth order, sibship size, childhood socioeconomic factors, perinatal characteristics, and Oral Health-Related Quality of Life and Periodontal Disease? Participants will simply have their routine periodontal examination, fill out the provided questionnaire, and continue their routine periodontal treatment.

DETAILED DESCRIPTION:
This study is planned to be carried out with 240 individuals between the ages of 18-30 who applied to Necmettin Erbakan University Faculty of Dentistry, Department of Periodontology for various reasons. In the Department of Periodontology, non-surgical periodontal treatment is performed for every patient diagnosed with periodontal disease after clinical and radiological evaluation.

Individual selection If there are patients who come to the Periodontology clinical secretariat for periodontal treatment and meet the inclusion criteria of the study, patients who agree to fill out the Oral Health Impact Profile-14 (OHIP-14) scales and the sociodemographic questionnaire including the number of siblings, sibling rankings, and other information about birth before the treatment and those who sign the consent form will be included in the study.

This study is actually a prospective survey study. In the study, researchers will ask patients who have undergone routine periodontal examinations by physicians in the clinic and who are planning for treatment to fill out questionnaires beforehand. Survey tracking will continue until the number of people filling out the survey is completed. After filling out the questionnaires, the routine non-surgical periodontal treatments of the patients will be continued.

Routine Periodontal Examination Routine periodontal examination will be used to measure plaque score, gingival score, pocket depths, and attachment loss. The amount of plaque; According to the plaque index (PI) defined by Silness and Löe, 0: no plaque; 1: the presence of plaque coming to the end of the end; 2: the presence of plaque visible; 3: will be considered as excessive plaque accumulation. Gingival index: As defined by Leue and Silness, 0: healthy gingiva; 1: there is slight inflammation and discoloration, there is no bleeding on probing, 2: there is moderate inflammation, hyperemia, bleeding on probing; 3: severe inflammation, hyperemia, ulceration, edema, spontaneous bleeding.

Patients will be diagnosed according to the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. Clinic gingival health would be defined as ≤3 mm probing depth and < 10% bleeding site. Participants will be diagnosed with periodontitis if interdental clinical attachment loss(CAL) is detected in 2 ≥2 adjacent teeth or if more than 3 mm buccal or oral CAL is detected in ≥2 teeth with a probing depth of ≥3 mm. The degree of periodontitis described will be based on the stage and grade system. For the definition of the four stages, the interdental CAL at the site of the greatest loss will be used. Stage classifies the severity and complexity of periodontitis (Stage I-II-III-IV), while grade is used to predict the likelihood of case progression (Grade A, B, C).

Periodontal probing depth and CAL will be evaluated at six sites per tooth. For pocket depth (PD) measurement with a periodontal probe, the probe will be placed parallel to the vertical axis of the tooth to reach the deepest point of the pocket, and the distance between the base of the pocket and the gingival edge will be manually recorded at the nearest millimeter mark. Similarly, the CAL will be measured as the distance between the enamel cementum boundary and the bottom of the pocket and recorded manually. When measuring CAL, at points where the enamel cementum boundary is not visible, it will be identified by tactile sense.

Scales to be applied:

Each patient participating in the study will be asked to fill out a questionnaire in which their birth and infancy conditions, childhood sociodemographic status, number and age of siblings, current sociodemographic status, and tooth brushing habits are specified. In addition, they will be asked to fill out the Oral Health Impact Profile-14 (OHIP-14).

When evaluating the age difference with the mother, under the age of 20 will be considered as very young, and 35 and over will be considered as advanced age. The age difference with the father will be stated as 24 and under. The following ranges will be used when assessing birth weight: <2500; 2500-3499; 3400- 3999; ≥4000.

Oral Health Impact Profile-14 (OHIP-14) OHIP-14 scale will be applied to the participants to determine Oral Health Related Quality of Life (OHRQoL). The total score of the responses on the OHIP-14 scale ranged from 0-56. Higher scores indicate a poorer quality of life. Any score higher than 14 will be taken as an indication of poor OHRQoL. The OHIP-14 questionnaire was translated into Turkish and its validity and reliability were made.

Statistical analysis Performed with the G Power program (G * Power 3.1 software; Heinrich Heine University, Düsseldorf, Germany) Correlation: According to the results of the power analysis for the Bivariate Normal Model, it was determined that 200 samples were appropriate when the critical correlation value was 0.3 at 0.90 power (1-β) with α (margin of error) = 0.05. However, assuming that 20% of patients quit, the study is planned to be conducted with a total of 240 people.

The data will be analyzed using the SPSS 11.0 statistical package (SPSS Inc., Chicago, USA). The chi-square test will be used to investigate the relationships between qualitative variables, the t-test will be used to compare two groups in terms of quantitative variables, and one-way ANOVA will be used to compare more than two groups in terms of quantitative variables. Pearson correlation analysis will be used for the relationship between qualitative variables. A p-value of 0.05 will be considered significant. Logistic regression analyses will be used to assess the roles of sibling size, birth order, and socioeconomic status in tooth loss and periodontal disease risk, and to control for potential confounders.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers between the ages of 18-30
* Not having any additional comorbidities
* Having at least 20 teeth in the entire mouth
* Getting diagnosed with healthy gums or Periodontitis
* Having spent his childhood with both parents
* Having at least 1 and at most 3 siblings

Exclusion Criteria:

* Being outside the inclusion criteria
* Not agreeing to participate in the study
* Having a psychiatric, mental or physical disability
* Being pregnant and lactating
* Having used any antibiotic, anti-inflammatory or any other drug that may affect - Smoking

Ages: 18 Years to 30 Years | Sex: All
Age Groups: Adult
Study Population: Patients who came to the Periodontology clinic secretariat for periodontal treatment and who met the inclusion criteria of the study will be included in the study. In order to minimize the effects of aging, the participant age was limited to 18-30. Only people whose parents were still married and who had a maximum of 3 siblings other than themselves were included in the study. It was thought that including participants whose parents were not currently married, whose parents were deceased, who had a half-sibling or who had more than three siblings would increase the confounding variables resulting from divorce or growing up in a family with multiple siblings, so these cases were not included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
socio demographic questionnaire and clinical parameters | Through study completion, an average of 4 months
  It will be determined whether there is a relationship between the current periodontal status of the participants and their birth order.
socio demographic and oral oral hygiene habits questionnaire | Through study completion, an average of 4 months
  It will be determined whether there is a relationship between the current oral hygiene habits of the participants and their birth order.
Oral Health Impact Profile-14 (OHIP-14) | Through study completion, an average of 4 months
  It will be determined whether there is a relationship between the current oral health related quality of life of the participants and their birth order. A high score of OHIP-14 indicates low OHRQoL.

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University, Konya, Konya/meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tastan Eroglu Z, Ozkan Sen D, Babayigit O, Yildiz K. Birth order, daycare attendance, and childhood socioeconomic status in relation to gingivitis: a cross-sectional study in Turkish young adults. BMC Oral Health. 2024 Nov 21;24(1):1420. doi: 10.1186/s12903-024-05215-4. PMID 39574099